CLINICAL TRIAL: NCT06047730
Title: Clinical Effect Evaluation of Laparoscopic Surgery for Ovarian Benign Tumors by Different Approaches
Status: Completed | Type: Observational
Sponsor: Yingchun Ma (Other)
Responsible Party: Sponsor-Investigator, Yingchun Ma, Clinical Effect Evaluation of Laparoscopic Surgery for Ovarian Benign Tumors by Different Approaches, Qianfoshan Hospital
Organization: Qianfoshan Hospital (Other)
Other Study IDs: V50KFC
Record Dates: First submitted 2023-09-14; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Laparoscope; Malignant Ovarian Tumor; Single-site Surgery
Keywords: Transumbilical laparoendoscopic single-site surgery,Giant malignant ovarian tumor
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- multi-port laparoscopic surgery
  Interventions: Procedure: operation ways
- transumbilical laparoendoscopic single-site surgery
  Interventions: Procedure: operation ways
- vaginal natural orifice transluminal endoscopic surgery
  Interventions: Procedure: operation ways

INTERVENTIONS:
Procedure: operation ways — nothing

SUMMARY:
Main purpose: To compare the intraoperative and postoperative recovery of laparoscopic surgery for ovarian benign tumors through different approaches; Secondary objective: Will vNOTES increase the risk of cesarean section during pregnancy and affect the quality of sexual life after surgery.

ELIGIBILITY:
Inclusion Criteria:

Preoperative consideration was for benign ovarian tumors requiring surgical treatment.

Exclusion Criteria:

* (1) Ovarian malignant tumor or borderline tumor was considered before surgery or proved during surgery. (2) Severe endometriosis, previous severe pelvic inflammation, peritonitis, and other serious pelvic adhesions are considered. (3) Pregnancy status. (4) Postoperative follow-up is not convenient and lost visitors.

Ages: 10 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: nothing
Sampling Method: Non-Probability Sample
Enrollment: 173 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
peroperative bleeding | during the operation time
  peroperative bleeding

SECONDARY OUTCOMES:
postoperative exhaust time | within 3 days after operation
  postoperative exhaust time

CONTACTS AND LOCATIONS:
Locations (1):
- Qianfoshan Hospital, The First Hospital affiliated of Shandong First Medical University, Jinan, Shandong, China